CLINICAL TRIAL: NCT03449927
Title: A Pilot Study of Implementation of a Nutritional Tool During Melphalan Autologous Transplant to Improve Caloric and Protein Intake
Brief Title: Implementation of a Nutritional Tool During Melphalan Autologous Transplant to Improve Caloric and Protein Intake
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 201711044
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Melphalan Autologous Transplant
Keywords: Nutrition Tool; Melphalan Autologous Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: Regular menu (Active Comparator): * Calorie count initiated on day +1 of transplant and ending upon count recovery
  * Symptom worksheet initiated on day +1 of transplant and ending upon count recovery (absolute neutrophil count of 1000)
  * Goals to monitor: calorie and protein intake, self-reported diarrhea and nausea
  * Interventions provided for control group: standard of care, verbal or printed handouts, standard educations created by Barnes Jewish Hospital (BJH) oncology dietitians
  Interventions: Other: Standard of care menu; Other: Self report dietary intake worksheet; Other: Post study questionnaire
- Intervention Arm: Specialized Menu (Experimental): * Calorie count and tool provided on day +1 and ending upon count recovery
  * Symptom worksheet initiated on day +1 of transplant and ending upon count recovery (absolute neutrophil count of 1000)
  * Goals to monitor: calorie and protein intake, self-reported diarrhea and nausea
  * Interventions provided for intervention group: standard of care provided by BJH oncology dietitians, tools including nausea and diarrhea menus and follow up by registered dietitian (RD) to provide additional counseling on menus as symptoms arise
  Interventions: Other: Specialized menu; Other: Self report dietary intake worksheet; Other: Post study questionnaire

INTERVENTIONS:
Other: Specialized menu — -Specialized menu that will guide participant food choices if the participant experiences nausea or diarrhea
  Arms: Intervention Arm: Specialized Menu
Other: Standard of care menu — -Standard registered dietitian support
  Arms: Control Arm: Regular menu
Other: Self report dietary intake worksheet — -Self report nausea and diarrhea
Other: Post study questionnaire — -Completed upon count recovery and prior to discharge

SUMMARY:
The purpose of this pilot before and after interventional study is to determine if early intervention and provision of menus regarding appropriate diet choices for melphalan autologous transplant patients experiencing nausea and diarrhea will improve nutrition status and overall calorie and protein intake throughout the transplant process.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing melphalan autologous transplants will be included in this study
* All patients that will be included in this pilot before and after interventional study will be inpatient on floors 5900, 6900 or 8900 of Barnes-Jewish Hospital
* Per hospital protocol, all patients who will receive a melphalan autologous transplant will be admitted and remain inpatient for the duration of the transplant process. There will be no exclusion for dietary restrictions or food allergies as the foodservice provided to patients is room service, all food allergies are noted and suitable alternatives are provided as a standard of service.
* Once a patient has been determined to meet criteria for the study, they will be approached by a member of the research team between day -2 and day 0 of transplant for consent. Patients must consent for the study by day +1 of transplant to be enrolled.

Exclusion Criteria:

* Patients <18 years of age
* Pregnant women
* Prisoners
* Patient unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Pre and post intervention mean total caloric intake | Through count recovery (10 days)
Mean total protein intake | Through count recovery (10 days)

SECONDARY OUTCOMES:
Mean daily caloric intake | Through count recovery (10 days)
Mean daily protein intake | Through count recovery (10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Stockmann, MS, RD, LD, Principal Investigator — Washington University School of Medicine; Meaghan Ryan, MSN, FNP-BC, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu